CLINICAL TRIAL: NCT05368714
Title: Suubi4StrongerFamilies: Addressing Child Behavioral Health by Strengthening Financial Stability and Parenting Among Families in Uganda
Brief Title: Suubi4StrongerFamilies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Fred Ssewamala, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01MH128905 (NIH); R01MH128905 (NIH)
Record Dates: First submitted 2022-05-01; First posted 2022-05-10 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Child Behavioral Health
Keywords: children; adolescents; child behavior; disruptive behaviors
MeSH Terms: conditions — Child Behavior; Problem Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three study conditions: 1) economic empowerment (EE) only, 2) multiple family group-based family strengthening (MFG-based FS), 3) combined EE+MFG-based FS.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Economic Empowerment (EE) (Experimental): EE consists of a child development account (CDA) held in the child's name in a financial institution registered by the Central Bank (Bank of Uganda).
  Interventions: Behavioral: Economic Empowerment (EE)
- Multiple Family Group (MFG) - based Family Strengthening (FS) Intervention: (Experimental): MFG-based consists of 16 sessions focused on building support for parents and families by providing opportunities for parents and children to communicate in a safe setting with other families who have shared experiences. Core components of MFG are known as 4Rs and 2S's: rules, responsibility, relationships, respectful communication, stress and social support.
  Interventions: Behavioral: Multiple Family Group based Family Strengthening (MFG-based FS)
- Combined EE plus MFG-based FS (Experimental): EE+ MFG-based FS combines both the child development account and 16 sessions of MFG.
  Interventions: Behavioral: EE plus MFG-based FS

INTERVENTIONS:
Behavioral: Economic Empowerment (EE) — EE will be provided via a child development account (CDA). CDAs provide children with basic financial education, introduce them to formal financial institutions, and incentivize them to save by matching their deposits. Any of the child's family members, relatives, or friends will be allowed and encouraged to contribute towards the CDA. The account will be matched with money from the program. The maximum family contribution to be matched by the program will be an equivalent of US $10 per month per family or US $120 for the 12-month intervention period.
  Arms: Economic Empowerment (EE)
Behavioral: Multiple Family Group based Family Strengthening (MFG-based FS) — MFG-based FS approach is a family-centered, group delivered, evidence-informed, strength-based intervention designed for children and adolescents whose families struggle with poverty and associated stressors. MFG is based on building support for parents and families by providing opportunities for parents and children to communicate in a safe setting with other families who have shared experiences. The core components of MFG are known as 4Rs and 2S's: rules, responsibility, relationships, respectful communication, stress and social support. Participants in this study arm will receive 16 session of MFG-based FS sessions, delivered by delivered by trained Community Health Workers and Parent Peers.
  Arms: Multiple Family Group (MFG) - based Family Strengthening (FS) Intervention:
Behavioral: EE plus MFG-based FS — EE plus MFG-based FS directly addresses both the economic needs and mental health functioning. It will consists of an EE intervention that comprises a family monetary savings program using CDAs, and a family-based dialogue and training via MFG focused on strengthening family relationships and mental health challenges.
  Arms: Combined EE plus MFG-based FS

SUMMARY:
The study will examine the mechanisms by which Economic Empowerment (EE) and Family Strengthening (FS) interventions targeting social, familial and context-specific drivers affect childhood behavioral health (CBH). The study will randomly assign 900 children in mid-upper primary school (10 to 14 years) to one of the three study arms (10 schools each): 1) EE only (n=300), 2) Multiple Family Group (MFG)-based FS only (n=300), and 3) combined EE+MFG-based FS (n=300). The interventions will be provided for 12 months. Assessments will occur at baseline, 12, 24 and 36 months.

DETAILED DESCRIPTION:
Children in Sub-Saharan Africa (SSA) are burdened by significant unmet mental health needs, with prevalence rates higher than 20%. The high rates of poverty, food insecurity, stigma and an inadequate health safety net system exacerbate serious childhood behavioral health (CBH) needs and impede an effective response. Youth disruptive behavioral disorders (DBDs) are a particularly serious concern as they persist through adolescence and adulthood. DBDs are also highly related to poor physical health and interpersonal challenges in adulthood. There is a need to address the context-specific social influences on CBH. Moreover, if children's needs are to be met in SSA, then: 1) implementing interventions designed and tested in SSA, and which mobilize resources within existing child-focused institutions (families, schools) is critical; 2) combined interventions that simultaneously target SSA-specific influences on CBH (family financial stability, culturally-based parenting), and can be delivered in collaboration with child/family-serving community settings (schools, faith-based and financial institutions) are necessary; and 3) group, community and population approaches to CBH are needed to drive scalable solutions.

This study will test the impact of Economic Empowerment (EE) and Family Strengthening (FS) interventions on childhood behavioral health. The study will utilize a longitudinal design with three active study conditions across 30 cluster-randomized primary schools to compare single and combination intervention options. The three study conditions are: 1) EE only, 2) MFG-based FS only, 3) combined EE+MFG-based FS. The interventions will be provided for 12 months; and assessments will occur at baseline, 12, 24 and 36 months.

The study will be guided by the following specific aims:

Aim 1: Examine the impact of EE only, MFG-based FS only, and combined EE+MFG-based FS on children's DBD symptoms and behavioral functioning;

Aim 2: Test the influence of EE only, MFG-based FS only, and combined EE+MFG-based FS on family financial stability (e.g., food and housing stability, material assets, savings), parenting and protective family processes (e.g., family organization, caregiver/child interaction, cohesion, support) and perceptions related to help-seeking (e.g., stigma) on CBH and functioning; and assess whether these change mechanisms mediate intervention effects on DBD symptoms and behavioral functioning, and explore moderation by context-specific moderators of intervention effects;

Aim 3: Qualitatively examine participants' experiences with each intervention arm.

ELIGIBILITY:
Inclusion criteria for children:

* Child in upper primary 5-7 (10 to 14 years)
* Meeting criteria for Opposition Defiant Disorder (ODD) or Conduct Disorder (CD)
* Willing to assent;

Inclusion criteria for caregivers:

* Adult caregiver of the child willing to consent
* Available for research and intervention activities.

Exclusion criteria:

-Inability to understand study procedures and participant rights as assessed during the informed consent/assent process with the child or parent. If the child or adult caregiver presents with emergency needs (e.g., hospitalization), needed care will be secured, rather than study participation.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 967 (Actual)
Dates: Start 2022-06-14 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in oppositional defiant disorder symptoms (reported by guardian) | Baseline, 12 months, 24 months, 36 months
  Change in oppositional defiant disorder symptoms will be measured using Iowa Conners scale. The scale has 16 items, with a score of 6 or higher on items 6-10 signifying positive oppositional disorder.
Change in impairment (reported by guardian) | Baseline, 12 months, 24 months, 36 months
  Change in child impairment impairment will be measured using the impairment scale. The scale has 7 items. A score of 3 or higher in any 4 or more items is considered a significant impairment.

SECONDARY OUTCOMES:
Change in child depression symptoms | Baseline, 12 months, 24 months, 36 months
  Change in child depression will be measured using the Child Depression Inventory. The study will measure the mean score on the CDI scale over time. The total score range between 0 and 28 with a high score indicating higher levels of depressive symptoms.
Change in Child Post Traumatic Stress Disorder (PTSD) symptoms | Baseline, 12 months, 24 months, 36 months
  Post traumatic stress will be measured using the Child PTSD reaction index. The study will measure the mean score on the Child PTSD Reaction Scale over time. The total score range between 0 and 120, with a high score indicating higher levels of PTSD.
Change in self concept | Baseline, 12 months, 24 months, 36 months
  Self concept will be measured using the Tennessee self-concept scale. The study will measure the mean score on the TSCS over time. The total score range between 20 and 100 with a high score indicating higher levels of self-concept.
Change in Family relations | Baseline, 12 months, 24 months, 36 months
  Family relations will be measured using items adapted from the family environmental scale and Family assessment scale. The study will measure the mean score over time, with higher scores indicating high levels of family relations/cohesion.
Change in Social Support | Baseline, 12 months, 24 months, 36 months
  Social Support from family members and friends will be measured using the social support behaviors scale. The study will measure the mean score over time. The total score range between 45- 225, with a higher score indicating high social support levels.
Change in Family stability | Baseline, 12 months, 24 months, 36 months
  Family stability will be assessed by asking respondents to indicate how long they have lived with their current family.
Change in mental health-related stigma | Baseline, 12 months, 24 months, 36 months
  Mental health-related stigma will be measured using the pediatric self-stigmatization scale. The study will measure mean scores over time. The total score range between 13 -52, with higher scores indicating high levels of mental health-related stigma.
Change in hopelessness symptoms | Baseline, 12 months, 24 months, 36 months
  Hopelessness will be measured using the Beck Hopelessness Scale. The study will assess the mean scores over time. The total score range between 0 - 20, with a higher score indicating higher levels of child hopelessness.
Change in Self Esteem | Baseline, 12 months, 24 months, 36 months
  Self esteem will be measured using Rosenberg Self-Esteem Scale. The study will assess the mean scores over time. The total score range between10 - 40, with a higher score indicating high levels of child self esteem.
Change in food insecurity and assets | Baseline, 12 months, 24 months, 36 months
  This will be measured using Household Food Insecurity Scale and Asset ownership. Total mean scores of both scales will be measured over time with a range of 0-25 and 0-21 respectively. A higher score indicates high levels of food security, economic stability and assets ownership.
Change in Access to services | Baseline, 12 months, 24 months, 36 months
  The study will measure the change in access to medical services as well as barriers to medical services over time.
Change in Savings | Baseline, 12 months, 24 months, 36 months
  Savings will be measured using official bank records/ monthly bank statements from the Child Development Accounts
Change in Perceived Social Support | Baseline, 12 months, 24 months, 36 months
  Perceived support from family members, friends and other individual will be measured using the Multidimensional Scale of Perceived Social Support. The study will measure the mean score on the MSPSS over time. The scale range between 12-84, with a higher score indicating high levels of perceived social support.

CONTACTS AND LOCATIONS:
Locations (1):
- International Center for Child Health and Development, Masaka, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Once all of the data has been de-identified, cleaned, and validated, and main findings have been published, the Investigators expect to share data with the scientific community. The research team will make datasets available to any individual who makes a direct request to the PI and indicates the data will be used for the purposes of research (per Code of Federal Regulations Title 45 Part 46: "Research is defined as a systematic investigation, including research development, testing and evaluation, designed to develop or contribute to generalizable knowledge."). In sharing participant data, the team will follow Washington University in St. Louis' Office of SponsoredProjects' data sharing agreement.
Supporting Information: Study Protocol, Analytic Code